CLINICAL TRIAL: NCT01970293
Title: AA Linkage for Alcohol Abusing Women Leaving Jail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1R01AA021732-01A1 (NIH)
Record Dates: First submitted 2013-08-08; First posted 2013-10-28 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Alcohol Use; AA Attendance; Sexual Risk Behavior
Keywords: Alcohol use; STI; Incarcerated women; AA
MeSH Terms: conditions — Alcohol Drinking; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Introduction to AA volunteer (Other)
  Interventions: Other: Introduction to AA volunteer
- AA materials offered (No Intervention)

INTERVENTIONS:
Other: Introduction to AA volunteer — In-person, in jail introduction to an AA volunteer, who will offer assistance in attending 2 AA meetings.
  Arms: Introduction to AA volunteer

SUMMARY:
The primary aims of this study are to test the hypotheses that among alcohol abusing and dependent jailed women returning to the community, adding an Alcoholic Anonymous (AA) linkage intervention will result in less alcohol use at follow-up, increased AA attendance once released, and decreased HIV/STI sexual risk behavior. Additionally, this study seeks to test the hypotheses that increased AA attendance will mediate the effect of the AA linkage intervention on alcohol use and that percent days abstinent will mediate the effect of the intervention on HIV/STI sexual risk-taking outcomes.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study participants must:

1. Be 18 years or older
2. Live in RI or MA within 20 miles of Providence and plan to remain in the area for the next 6 months
3. Meet DSM-IV criteria for alcohol abuse or dependence in the last six months
4. Do not expect to attend residential alcohol or drug treatment upon release
5. Report STI/HIV sexual risk defined as unprotected heterosexual sex at least three times in the three months prior to incarceration
6. Speak English.
7. Be currently held at the Rhode Island Adult Correctional Institutions Jail facility

Women will be excluded from participation if they:

1. Cannot provide the name of at least two locator persons who will know where they can be found.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Change in number of alcohol use days from baseline to 6 months | Baseline, 1, 3, and 6 months
  Timeline Followback (TLFB) participant recall of alcohol use days.

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Timko C, Chatav Schonbrun Y, Anderson B, Johnson JE, Stein M. Perceived Substance Use Norms Among Jailed Women with Alcohol Use Disorders. Alcohol Clin Exp Res. 2020 Sep;44(9):1834-1841. doi: 10.1111/acer.14403. Epub 2020 Sep 2. PMID 32876998
- [Derived] Schonbrun YC, Kurth M, Johnson J, Timko C, Stein M. Participant Evaluation of Twelve-Step Group Linkage for Jailed Women With Alcohol Use Disorder. Int J Offender Ther Comp Criminol. 2019 Mar;63(4):610-623. doi: 10.1177/0306624X18805598. Epub 2018 Oct 12. PMID 30311822
- [Derived] Timko C, Johnson JE, Kurth M, Schonbrun YC, Anderson BJ, Stein MD. Health Services Use Among Jailed Women with Alcohol Use Disorders. J Behav Health Serv Res. 2019 Jan;46(1):116-128. doi: 10.1007/s11414-018-9634-7. PMID 30238292
- [Derived] Hailemariam M, Stein M, Anderson B, Schonbrun YC, Moore K, Kurth M, Richie F, Johnson JE. Correlates of alcoholics anonymous affiliation among justice-involved women. BMC Womens Health. 2018 Jul 11;18(1):125. doi: 10.1186/s12905-018-0614-0. PMID 29996829